CLINICAL TRIAL: NCT02336529
Title: Tenderpoint and Ultrasound Guided Nerveblocks for Persistent Pain After Breast Cancer Surgery
Brief Title: Nerveblocks for Persistent Pain After Breast Cancer Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kenneth Geving Andersen (Other)
Responsible Party: Sponsor-Investigator, Kenneth Geving Andersen, Research fellow, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: H-3-2013-172
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Pain; Neuropathic Pain; Breast Cancer
Keywords: postoperative
MeSH Terms: conditions — Pain; Neuralgia; Breast Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ICBN, active (Experimental): Ultrasound guided injection of bupivacain, 10mL, 0.5% in proximity of the ICBN
  Interventions: Drug: Bupivacaine
- ICBN, placebo (Placebo Comparator): Ultrasound guided injection of NaCl, 10mL in proximity of the ICBN
  Interventions: Drug: NaCl
- Tenderpoint, active (Experimental): Ultrasound guided injection of bupivacain, 20mL, 0.25% in the tenderpoint
  Interventions: Drug: Bupivacaine
- Tenderpoint, placebo (Placebo Comparator): Ultrasound guided injection of NaCl, 20mL in the tenderpoint
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Bupivacaine
  Arms: ICBN, active; Tenderpoint, active
Drug: NaCl
  Arms: ICBN, placebo; Tenderpoint, placebo

SUMMARY:
Persistent pain after breast cancer surgery (PPBCS) affects 25-60% of breast cancer survivors and nerve damage has been implicated as the cause of this neuropathic pain condition. Local anaesthetic blockade of tenderpoints and the intercostobrachial nerve (ICBN) could provide clues to pathophysiological mechanisms as well as aiding diagnosis and treatment of PPBCS but has never been attempted. The aims of this study is to examine clinical effect of ultrasound guided blockades of the ICBN and tenderpoints of pain.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 year after surgery for breast cancer
* Women aged 18 or over
* Suffering from persistent pain in the breast, side of chest, axilla or arm (NRS 4 or over)

Exclusion Criteria:

* Previous cosmetic surgery
* bilateral cancer
* pregnant or lactating
* other disease in the nervous system
* in treatment for psychiatric disease
* unable to understand Danish
* unable to give informed concent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Summed pain intensity | At least 1 year after surgery
  The summed pain intensity (of pain at rest (0-10), pain during movement (0-10) and pressure pain (at 100kPa in point of maximum pain) (0-10)) 0-30

SECONDARY OUTCOMES:
Pain at rest, pain during movement and pressure pain | At least 1 year after surgery
  Pain intensity of pain at rest (0-10), pain during movement (0-10) and pressure pain (at 100kPa in point of maximum pain) (0-10)
Pain related reduction of physical function | At least 1 year after surgery
  Reduction of physical function

CONTACTS AND LOCATIONS:
Overall Officials: Nelun Wijayasinghe, MD, Principal Investigator — Rigshospitalet, University of Copenhagen; Kenneth G Andersen, MD, PhD, Study Chair — Rigshospitalet, University of Copenhagen

REFERENCES:
- [Background] Wijayasinghe N, Andersen KG, Kehlet H. Neural blockade for persistent pain after breast cancer surgery. Reg Anesth Pain Med. 2014 Jul-Aug;39(4):272-8. doi: 10.1097/AAP.0000000000000101. PMID 24918332